CLINICAL TRIAL: NCT00866229
Title: Efficacy and Adverse Effect of Simvastatin Compare to Rosuvastatin in SLE Patients With Corticosteroid Therapy and High LDL Cholesterol Level
Brief Title: Efficacy and Adverse Effect of Simvastatin Compare to Rosuvastatin in Systemic Lupus Erythematosus (SLE) Patients With Corticosteroid Therapy and High Low-Density Lipoprotein (LDL) Cholesterol Level
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramathibodi Hospital (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Parawee Suwannalai , M.D., Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID03-51-15
Record Dates: First submitted 2009-03-19; First posted 2009-03-20 (Estimated); Last update posted 2009-03-20 (Estimated); Status verified 2009-03

CONDITIONS: Systemic Lupus Erythematosus; High LDL Cholesterol Level
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Rosuvastatin Calcium; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Rosuvastatin — 10 mg per day for 12 weeks
Drug: Simvastatin — 20 mg per day

SUMMARY:
Early statin therapy in SLE patients that have high cholesterol level and other atherosclerosis risk should reduce atherosclerosis and coronary artery events in later course of disease. By the way, statin is used in restricted groups of rheumatologists due to awareness of side effects; myositis and hepatitis, that are frequently found in SLE patients more so than other groups of atherosclerosis patients and reporting data of autoimmune diseases that occur after statin use.

ELIGIBILITY:
Inclusion Criteria:

* SLE patients that on prednisolone more than 30 mg/day
* Normal liver faction: AST and ALT < 80 mg/dl
* Normal muscle enzyme : CPK < 100 U/L
* LDL cholesterol level > 100 mg/dl

Exclusion Criteria:

* Patients that was treated with pulse methylprednisolone or corticosteroid equivalent to prednisolone > 1mg/kg/day at screening.
* Statin allergy
* On statin treatment before screening
* On cyclosporine, antifugal (azole group), antibiotics (macrolide group), rifampicin, warfarin, phenytoin
* Pregnancy
* Abnormal liver function: AST or ALT > 80 mg/dl
* Abnormal muscle enzyme : CPK > 300 U/L

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2008-04; Primary Completion 2010-03 (Estimated); Study Completion 2010-06 (Estimated)

PRIMARY OUTCOMES:
Percentage reduction of LDL Cholesterol level | 6 and 12 weeks

SECONDARY OUTCOMES:
Proportion of patients that have transminitis, myositis or active SLE | 6,12, 18 and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Parawee Suwannalai, M.D., Principal Investigator — Ramathibodi Hospital
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Bangkok, Thailand